CLINICAL TRIAL: NCT04192838
Title: Long-term Outcomes and Quality of Life of Incisional Ventral Hernia Repair by Open or Laparoscopy Surgery: Randomized Clinical Trial Extension
Brief Title: Incisional Hernia Repair Long-term Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Salvador Peiro (Other)
Responsible Party: Sponsor-Investigator, Salvador Peiro, Head of Health Services Department, Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana
Organization: Fundación para el Fomento de la Investigación Sanitaria y Biomédica de la Comunitat Valenciana (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IH/AV/2017
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Incisional Hernia
Keywords: Incisional hernia; Laparoscopic surgery; Recurrence; Health Related Quality of Life
MeSH Terms: conditions — Incisional Hernia; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LVHR (Experimental): Laparoscopic incisional ventral hernia repair
  Interventions: Procedure: Laparoscopic incisional ventral hernia repair
- OVHR (Active Comparator): Open incisional ventral hernia repair
  Interventions: Procedure: Open incisional ventral hernia repair

INTERVENTIONS:
Procedure: Laparoscopic incisional ventral hernia repair — Laparoscopic repair of incisional ventral hernias (5-15 cm) with adouble-layer polypropylene- expanded polytetrafluoroethylene (ePTFE) mesh.
  Arms: LVHR
Procedure: Open incisional ventral hernia repair — Standard polypropylene mesh was positioned as an inlay, or as an onlay over the external oblique fascia (i.e., subcutaneously), as preferred by the operating team. The mesh was fixed with absorbable stitches. Drains were usually placed.
  Arms: OVHR

SUMMARY:
Long-term extension of a previous trial comparing outcomes after open (OVHR) or laparoscopic incisional ventral hernia repair (LVHR), assessing recurrence, reoperation, intraperitoneal mesh-related complications and self-reported quality-of-life with 10-15 years of follow-up.

DETAILED DESCRIPTION:
Long-term studies comparing outcomes after open (OVHR) or laparoscopic incisional ventral hernia repair (LVHR) are scarce. We carried-out a long-term extension of a previous trial comparing both approaches, assessing recurrence, reoperation, intraperitoneal mesh-related complications and self-reported quality-of-life with 10-15 years of follow-up.

Patients will be followed to assess recurrence (main endpoint), reoperation, mesh complications and death, from the date of index surgery (between 2003 to 2006) until recurrence, death or study completion with a clinical revision (between 2017 to 2019) whichever was first. By intention to treat, incidence rates of recurrence, reintervention and death by 1000 person-year of follow-up will be estimated, and also rates of mesh complications by 1000 person-year for the LVHR group excluding conversions. Quality of life, using the European Hernia Society Quality of Life score (EuraHS-QoL), will be assessed for survivors no reoperated patients

ELIGIBILITY:
Inclusion Criteria:

* Incisional hernia between 5 and 15 cm in largest diameter
* No ontraindication for laparoscopic surgery.

Exclusion Criteria:

* Patients with any type of stoma,
* Non-residente in the Valencia región

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2003-02-24 (Actual); Primary Completion 2019-12-24 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Hernia recurrence | 10-15 years
  Rate of participants with hernia recurrence assessed by: 1) clinical evaluation during the first year of follow-up, taking advantage of the original RTC data, available for all patients in the study; 2) clinical evaluation, accompanied when necessary by an abdominal CT scan, carried out between 2017 and 2019 for living patients who accepted participation in the extension study; 3) review of the EMR, including available abdominal CT scans close to patients' death, for patients deceased prior to the clinical evaluation of the extension study.

SECONDARY OUTCOMES:
Surgical repair of recurrent incisional hernia | 10-15 years
  Rate of participants with a hernia reoperation assessed by: 1) clinical evaluation during the first year of follow-up, taking advantage of the original RTC data, available for all patients in the study; 2) clinical evaluation carried out between 2017 and 2019 for living patients who accepted participation in the extension study; 3) review of the EMR for patients deceased prior to the clinical evaluation of the extension study.
Mesh related complications | 10-15 years
  Rate of participants with a reoperation for intestinal obstruction, or mesh extrusion, or intestinal fistulas, or adhesion syndrome treated conservatively. Only for intraperitoneal mesh
Health Related Quality of Life: EuraHS-QoL questionnaire | 10-15 years
  The EuraHS-QoL questionnaire was used for assessing HRQoL in living no reoperated patients who accepted participation in the clinical evaluation of the extension study. The EuraHS-QoL scale is a hernia specific HRQoL self-administered questionnaire with 9 items that can be scored by the patient in an 11-point scale (from 0 to 10). The total score ranges from 0-90, with the lower scores being the most favourable outcome.

OTHER OUTCOMES:
Rate of deaths | 10-15 years
  Death for any cause

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Asencio-Arana, MD, PhD, Principal Investigator — Arnau de Vilanova University Hospital
Locations (3):
- Spain (3):
  - Francesc de Borja Hospital, Gandia, Valencia
  - Lluis Alcanyis Hospital, Xàtiva, Valencia
  - Arnau de Vilanova Hospital, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Asencio F, Aguilo J, Peiro S, Carbo J, Ferri R, Caro F, Ahmad M. Open randomized clinical trial of laparoscopic versus open incisional hernia repair. Surg Endosc. 2009 Jul;23(7):1441-8. doi: 10.1007/s00464-008-0230-4. Epub 2008 Dec 31. PMID 19116750
- [Derived] Asencio F, Carbo J, Ferri R, Peiro S, Aguilo J, Torrijo I, Barber S, Canovas R, Andreu-Ballester JC. Laparoscopic Versus Open Incisional Hernia Repair: Long-Term Follow-up Results of a Randomized Clinical Trial. World J Surg. 2021 Sep;45(9):2734-2741. doi: 10.1007/s00268-021-06164-7. Epub 2021 May 20. PMID 34018042